CLINICAL TRIAL: NCT01024309
Title: A Prospective, Randomized, Clinical Trial Comparing the Clinical Outcomes Following Total Hip Arthroplasty by a Single Surgeon Using Either a Mini-posterior Approach or a Direct Anterior Approach
Brief Title: A Trial Comparing Mini-posterior Approach and Direct Anterior Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09072
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Osteoarthritis
Keywords: total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mini-Posterior Approach (Active Comparator): Mini-Posterior surgical approach for total hip arthroplasty
  Interventions: Procedure: Mini-Posterior surgical approach for total hip arthroplasty
- Direct Anterior Approach (Experimental): Direct Anterior surgical approach for total hip arthroplasty
  Interventions: Procedure: Direct Anterior surgical approach for total hip arthroplasty

INTERVENTIONS:
Procedure: Mini-Posterior surgical approach for total hip arthroplasty — Mini-Posterior surgical approach for total hip arthroplasty
  Arms: Mini-Posterior Approach
Procedure: Direct Anterior surgical approach for total hip arthroplasty — Direct Anterior surgical approach for total hip arthroplasty
  Arms: Direct Anterior Approach

SUMMARY:
The purpose is to determine if differences exist in the attainment of functional milestones that reflect activities of daily living between mini-posterior and direct anterior approach total hip arthroplasty (THA). The investigators also hope to determine if the general health outcome after direct anterior total hip arthroplasty was better than that after mini-posterior-incision total hip arthroplasty as measured with Short Form-12 (SF-12) scores, and to evaluate variation of surgical factors of the two procedures on the basis of the operative time, component positioning, and occurrence of early complications.

DETAILED DESCRIPTION:
A number of studies have compared surgical approach for total hip arthroplasty. The influence of surgical outcome as a function of approach comparing mini-posterior to direct anterior has not been reported in a randomized, prospective manner.

Standard primary total hip arthroplasty (THA) can reliably alleviate pain, improve function, and improve the quality of life in a broad section of patients with end stage arthrosis of the hip. However, minimally invasive approaches, such as the direct anterior and mini-posterior approaches, have been devised with the goal of decreasing peri-operative pain, speed early postoperative function, and improve patient satisfaction with the procedure, compared with standard THA. These patient centered goals are combined with the surgeon's desire of a safe, reproducible minimally invasive procedure that has durable, properly positioned components.

There are currently no prospective, randomized studies comparing the direct anterior approach to total hip arthroplasty with other minimally invasive approaches. The mini-posterior approach has been studied extensively, with promising results. Others have compared the mini-posterior approach with other minimally invasive procedures, and at the current time, has the most prospective data demonstrating its superiority as a minimally invasive approach. Pagnano performed a prospective, randomized trial comparing the early clinical results of mini -posterior THA with Two-incision THA. The results found that the early attainment of functional milestones was shorter in the mini-posterior group.

The purpose is to determine if differences exist in the attainment of functional milestones that reflect activities of daily living between mini-posterior and direct anterior approach total hip arthroplasty (THA). The investigators also hope to determine if the general health outcome after direct anterior total hip arthroplasty was better than that after mini-posterior-incision total hip arthroplasty as measured with Short Form-12 (SF-12) scores, and to evaluate variation of surgical factors of the two procedures on the basis of the operative time, component positioning, and occurrence of early complications.

ELIGIBILITY:
Inclusion Criteria:

* The subject is willing and able to understand, sign and date the study specific Patient Informed Consent and Health Insurance Portability and Accountability Act (HIPPA) authorization to volunteer participation in the study.
* The subject is between 25 and 80 years of age at the time of surgery.
* The subject has elected to undergo primary total hip arthroplasty for osteoarthritis.
* The subject is psychosocially, mentally and physically able to comply with the requirements of the study including post-operative clinical, radiographic evaluations and completion of patient questionnaires.
* The subject is skeletally mature.

Exclusion Criteria:

* The subject has a BMI greater than 35.
* The subject has had a previous total hip arthroplasty.
* The subject has inflammatory arthritis.
* The subject has any type of infection.
* The subject has developmental dysplasia of the hip.
* The subject has a known metal allergy.
* The subject has an extreme offset of greater than 50 mm.
* The subject has an acetabular deformity requiring advanced reconstructive techniques.
* The subject has Charcot's disease.
* The subject has Paget's disease
* Dependence on narcotics for 6 months (or longer)

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Bohannon Mason, MD, Principal Investigator — OrthoCarolina, P.A.
Locations (1):
- OrthoCarolina, P.A., Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 66 volunteer participants were enrolled during routine clinical practice of the principal investigator between the dates of 12/8/2009 and 10/9/2012.
Pre-assignment Details: 12 patients withdrew participation prior to randomization
Period: Overall Study
Arm/Group | Mini-Posterior Approach | Direct Anterior Approach
Started | 35 | 31
Completed | 27 | 27
Not Completed | 8 | 4
Not completed — Physician Decision | 4 | 0
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mini-Posterior Approach | Direct Anterior Approach | Total
Number analyzed (Participants) | 35 | 31 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 17 | 14 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (9.4) | 63.4 (8.6) | 63.8 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 17 | 15 | 32
Region of Enrollment [Number; unit: participants]
  United States | 35 | 31 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Days for Discontinue Assistive Devices
Description: The primary early functional endpoint is the difference between groups in the postoperative days that patients require any assistive devices for ambulation. Lower number of days indicate better outcomes.
Time Frame: 6 week
Population: A total of 54 participants returned for follow-up at 6 weeks. The remaining patients did not return to the clinic for follow-up at 6 weeks.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Mini-Posterior Approach | Direct Anterior Approach
Number analyzed (Participants) | 27 | 27
days | 28 [20 to 42] | 22 [12 to 30]
Statistical Analysis 1: Comparison: Mini-Posterior Approach vs Direct Anterior Approach; Test type: Superiority or Other; p = .04, Wilcoxon (Mann-Whitney) — Apriori level of significance was 0.05; Wilcoxon Rank Sum was used

2. Secondary Outcome: Harris Hip Score
Description: The postoperative rate of improvement in functional outcome, measured by the Harris Hip Score (HHS). The HHS was developed to assess the results of hip surgery and is intended to evaluate various hip disabilities and methods of treatment in an adult population. The domains covered are pain, function, absence of deformity, and range of motion. The function domain consists of daily activities (stair use, using public transportation, sitting, and managing shoes and socks) and gait (limp, support needed, and walking distance). Deformity takes into account hip flexion, adduction, internal rotation, and extremity length discrepancy. Range of motion measures hip flexion, abduction, external and internal rotation, and adduction. There are 10 items, which are summed to create a score out of 100. The score has a range of 0 (wost possible outcome) to 100 (best possible outcome) covering pain (0-44 points), function (0-47 points), absence of deformity (4 points), and range of motion (5 points).
Time Frame: 3 week
Population: A total of 53 participants returned for follow-up at 3 weeks. The remaining patients did not return to the clinic for follow-up at 3 weeks.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Mini-Posterior Approach | Direct Anterior Approach
Number analyzed (Participants) | 27 | 26
units on a scale | 81 [74 to 89] | 86.5 [77 to 95]
Statistical Analysis 1: Comparison: Mini-Posterior Approach vs Direct Anterior Approach; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney) — the a priori threshold for statistical significance was 0.05; Wilcoxon Rank Sum Test

3. Secondary Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Description: Total score from the Western Ontario and McMaster Universities Arthritis Index (WOMAC), which is a widely used set of standardized questionnaires used to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. WOMAC measures five items for pain (score range 0-20), two for stiffness (range 0-8), and 17 for functional limitation (range 0-68). Physical functioning questions cover everyday activities such as stair use, standing up from a sitting or lying position, standing, bending, walking, getting in/out of a car, shopping, putting on or taking off socks, lying in bed, getting in or out of a bath, sitting, and heavy and light household duties. It produces three subscale scores (pain, stiffness, and physical function) and a total score. These scores are transformed into a scale of 0 (worst possible outcome) to 100 (best possible outcome) for ease of interpretation and comparison with other studies.
Time Frame: 3 week
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Mini-Posterior Approach | Direct Anterior Approach
Number analyzed (Participants) | 27 | 26
units on a scale | 91.48 [85.01 to 96.19] | 87.20 [74.92 to 92.03]
Statistical Analysis 1: Comparison: Mini-Posterior Approach vs Direct Anterior Approach; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney) — the a priori threshold for statistical significance was 0.05; Wilcoxon Rank Sum Test was used

4. Secondary Outcome: Abduction Angle
Description: Abduction angle is a radiographic measure of implant position. 40 degrees of abduction is optimal. 30-50 degrees of anteversion indicates correct placement of prosthetic joint. Values closer to 40 degrees indicate better placement.
Time Frame: 6 wk
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Mini-Posterior Approach | Direct Anterior Approach
Number analyzed (Participants) | 27 | 27
degrees | 40 [36 to 42] | 38 [36 to 41]
Statistical Analysis 1: Comparison: Mini-Posterior Approach vs Direct Anterior Approach; Test type: Superiority or Other; p = 0.22, Wilcoxon (Mann-Whitney) — the a priori threshold for statistical significance was 0.05; Wilcoxon Rank Sum Test was used

5. Secondary Outcome: Anteversion Angle
Description: Anteversion angle is a radiographic measure of implant position. 35 degrees of anteversion is optimal. 25-45 degrees of anteversion indicates correct placement of prosthetic joint. Values closer to 35 degrees indicate better placement.
Time Frame: 6 week
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Mini-Posterior Approach | Direct Anterior Approach
Number analyzed (Participants) | 27 | 27
degrees | 29 [26 to 32] | 26 [24 to 28]
Statistical Analysis 1: Comparison: Mini-Posterior Approach vs Direct Anterior Approach; Test type: Superiority or Other; p = .0029, Wilcoxon (Mann-Whitney) — the a priori threshold for statistical significance was 0.05; Wilcoxon Rank Sum Test was used

6. Secondary Outcome: Harris Hip Score
Description: as for outcome 2
Time Frame: 6 week
Population: 54 participants returned for follow-up at 6 weeks. A total of 5 participants did not complete the Harris Hip Score instrument in its entirety at this appointment and, thus, were excluded from the analysis. The remaining patients did not return to the clinic for follow-up at 6 weeks.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Mini-Posterior Approach | Direct Anterior Approach
Number analyzed (Participants) | 26 | 23
units on a scale | 93 [89 to 98] | 97 [90 to 98]
Statistical Analysis 1: Comparison: Mini-Posterior Approach vs Direct Anterior Approach; Test type: Superiority or Other; p = 0.13, Wilcoxon (Mann-Whitney) — the a priori threshold for statistical significance was 0.05; Wilcoxon Rank Sum Test was used

7. Secondary Outcome: WOMAC
Description: as for outcome 3
Time Frame: 6 week
Population: A total of 54 participants returned for follow-up at 6 weeks. 3 participants did not complete the WOMAC in its entirety at this appointment and, thus, were excluded from the analysis. The remaining patients did not return to the clinic for follow-up at 6 weeks.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Mini-Posterior Approach | Direct Anterior Approach
Number analyzed (Participants) | 25 | 26
units on a scale | 95.72 [91.48 to 98.92] | 95.41 [87.83 to 97.37]
Statistical Analysis 1: Comparison: Mini-Posterior Approach vs Direct Anterior Approach; Test type: Superiority or Other; p = 0.29, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance was 0.05; Wilcoxon Rank Sum

8. Secondary Outcome: Harris Hip Score
Description: as for outcome 2
Time Frame: 12 month
Population: A total of 37 participants returned for follow-up at 12 months. The remaining patients did not return to the clinic for follow-up at 12 months.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Mini-Posterior Approach | Direct Anterior Approach
Number analyzed (Participants) | 20 | 17
units on a scale | 97.5 [87 to 100] | 98 [94 to 100]
Statistical Analysis 1: Comparison: Mini-Posterior Approach vs Direct Anterior Approach; Test type: Superiority or Other; p = 0.23, Wilcoxon (Mann-Whitney) — the a priori threshold for statistical significance was 0.05; Wilcoxon Rank Sum Test was used

9. Secondary Outcome: WOMAC
Description: as for outcome 3
Time Frame: 12 month
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Mini-Posterior Approach | Direct Anterior Approach
Number analyzed (Participants) | 20 | 17
units on a scale | 97.37 [88.84 to 100] | 97.37 [92.07 to 99.46]
Statistical Analysis 1: Comparison: Mini-Posterior Approach vs Direct Anterior Approach; Test type: Superiority or Other; p = 0.49, Wilcoxon (Mann-Whitney) — the a priori threshold for statistical significance was 0.05; Wilcox Rank Sum Test

ADVERSE EVENTS:
Arm/Group | Mini-Posterior Approach | Direct Anterior Approach
Serious Adverse Events (participants affected / at risk) | 3/27 | 1/27
Other Adverse Events (participants affected / at risk) | 1/27 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mini-Posterior Approach (N=27) | Direct Anterior Approach (N=27)
Chest pain and tightness (Cardiac disorders) | 1 (1) | 0 (0) — Emergency Room Visit
Medication Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Emergency Room Visit
Superficial hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gallstone (Gastrointestinal disorders) | 1 (1) | 0 (0) — Surgery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mini-Posterior Approach (N=27) | Direct Anterior Approach (N=27)
Calcar bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dehydration and gastroenteritis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Surgical incision complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Capsular stitch popped

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No